CLINICAL TRIAL: NCT07117799
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 2 ARM, 2-PERIOD, CROSS-OVER, SINGLE-DOSE STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE RELATIVE BIOAVAILABILITY OF TWO PF-07248144 CLINICAL TRIAL FORMULATIONS
Brief Title: A Study to Learn About How Different Forms of Study Medicine PF-07248144 Are Taken Up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4551005
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adults
Keywords: Bioavailability; Bioequivalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-07248144 Form 1 (uncoated) Arm (Experimental): Period 1: Participants received Form 1 in a single dose of tablet fasted Period 2: Participants received Form 5 in a single dose of tablet fasted
  Interventions: Drug: PF-07248144
- PF-07248144 Form 5 (film-coated) Arm (Experimental): Period 1: Participants received Form 5 in a single dose of tablet fasted Period 2: Participants received Form 1 in a single dose of tablet fasted
  Interventions: Drug: PF-07248144
- PF-07248144 Form 5 (film-coated) Adaptive Arm (Experimental): Period 1: Fasted participants received a single dose of tablet of Form 1 orally Period 2: Participants received a single dose of tablet orally of Form 5 in a fed state
  Interventions: Drug: PF-07248144

INTERVENTIONS:
Drug: PF-07248144 — Period 1: Participants received Form 1 in a single dose of tablet fasted Period 2: Participants received Form 5 in a single dose of tablet fasted
Drug: PF-07248144 — Period 1: Participants received Form 5 in a single dose of tablet fasted Period 2: Participants received Form 1 in a single dose of tablet fasted
Drug: PF-07248144 — Period 1: Fasted participants received a single dose of tablet of Form 1 orally Period 2: Participants received a single dose of tablet orally of Form 5 in a fed state

SUMMARY:
Study has two arms. Arm 1 has two cohorts in which each cohort, under the fasted state, will either be given a single oral dose of Form 1 in Period 1 followed by a single oral dose of Form 5 in Period 2 or a single oral dose of Form 5 in Period 1 followed by a single oral dose of Form 1 in Period 2. A single oral dose of Form 1 will be administered in Arm 2 Period 1 under the fasted state. The results from Arm 1 will inform whether a different dose of Form 5 will be administered under the fasted state or if Form 5 will be administered under the fed state in Arm 2 Period 2.

ELIGIBILITY:
Inclusion Criteria

* Participants of nonchildbearing potential , inclusive, at screening, who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead electrocardiograms (ECGs).
* Body mass index (BMI) of 18-32 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria

* Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention
* Prior use of epigenetic modifying agents
* Current use of any prohibited concomitant medication(s) or unwillingness or inability to use a required concomitant medication(s)
* Additionally, current use or anticipated need for food or drugs that are known strong inducers or inhibitors of CYP2C9 or CYP3A4, including their administration within 14 days or 5 half-live of the strong inducers or inhibitors of CYP2C9 or CYP3A4, whichever is longer, prior to first dose of study intervention, during the treatment period, and within 2 days after the last dose of PF-07248144
* Proton pump inhibitors must be discontinued at least 5 days prior to the first dose of study medication and throughout treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-07248144 Form 1 uncoated tablet | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, and 168 hours post-dose
AUCinf for PF-07248144 Form 5 film-coated tablet | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, and 168 hours post-dose
Maximum Observed Plasma Concentration (Cmax) for PF-07248144 Form 1 uncoated tablet | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, and 168 hours post-dose
Cmax for PF-07248144 Form 5 film-coated tablet | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, and 168 hours post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment Related AEs and SAEs | From Baseline up to Day 35
Number of Participants With Laboratory Test Abnormalities | From Baseline up to Day 35
Number of Participants With Vital Signs Values Meeting Categorical Summarization Criteria | From Baseline up to Day 35
Number of Participants With Clinically Significant Physical Examination Abnormalities | From Baseline up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4551005